CLINICAL TRIAL: NCT07036523
Title: A Double-blind, Randomised, Placebo-controlled, Parallel Group, Phase IIa Trial to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of BI 765423 Administered Intravenously With or Without Standard of Care in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Find Out Whether BI 765423 Has an Effect on Lung Function in People With Idiopathic Pulmonary Fibrosis (IPF) With or Without Standard Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1493-0002; 2025-520658-12-00 (Registry Identifier: CTIS (EU)); U1111-1317-7542 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 765423 (Experimental)
  Interventions: Drug: BI 765423
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 765423 — BI 765423
  Arms: BI 765423
Drug: Placebo — Placebo to BI 765423
  Arms: Placebo

SUMMARY:
This study is open to adults who are at least 40 years old and have idiopathic pulmonary fibrosis (IPF). People can participate in the study if they have a forced vital capacity (FVC) greater than or equal to 45% of the predicted value and fibrosis of 20% or more confirmed by a high-resolution computed tomography (HRCT) scan. The purpose of this study is to find out if a medicine called BI 765423 can improve lung function in people with IPF. The study will compare BI 765423 with a placebo to see if there is a difference in lung capacity after 3 months of treatment and will also look at changes in certain markers related to lung health.

Participants are put into two groups randomly, which means by chance. One group receives the study medicine, and the other group receives a placebo. Placebo looks like BI 765423 but does not contain any study medicine. The study medicine is given as an infusion into a vein every four weeks.

Participants are in the study for 8-10 months. During the study, participants may continue their regular treatment for IPF. During the study they visit the study site several times for screening, treatment, and follow-up. Doctors regularly test lung function by measuring FVC and take blood samples to measure study endpoints. The results are compared between the two groups to see whether the treatment works. The doctors also check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria :

1. 40 years of age or older at the time of informed consent signature.
2. Signed and dated written informed consent in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
3. Male or female patients. Male patients with Woman of childbearing potential (WOCBP) sexual partners must use contraception (male condom) to avoid exposure via seminal fluid during treatment and for a specific period after last drug intake. Women can only be included if they are of non-childbearing potential, defined as meeting at least one of the below conditions:

   * Permanently surgically sterilised (hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy)
   * Postmenopausal, defined as no menses for 12 months without an alternative medical cause. In questionable cases of postmenopausal status:

     * Women not using sex hormone medication such as hormone replacement therapy may be included if a blood sample confirms levels of follicle stimulating hormone (FSH) > 40 U/L and estradiol < 30 ng/L"
4. Patients with a documented diagnosis of IPF prior to Visit 1, confirmed by the investigator as per the 2022 American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) Guideline and, if available, surgical lung biopsy or transbronchial lung cryobiopsy histopathology report.
5. Patients with a high-resolution computed tomography (HRCT) taken within 12 months of Visit 1 (or during the screening period, if not available) confirming "UIP" or "probable UIP" HRCT pattern consistent with the clinical diagnosis of IPF by central review (prior to Visit 2).

   * Patients with an "indeterminate" HRCT finding are eligible if a clinical diagnosis of IPF can be confirmed based on an historical histopathology report of a surgical lung biopsy or cryobiopsy demonstrating a "UIP" or "Probable UIP" pattern.
   * Patients with an "alternative diagnosis" HRCT finding are eligible if a clinical diagnosis of IPF can be confirmed based on an historical histopathology report of a surgical lung biopsy or cryobiopsy demonstrating a "UIP" pattern."
6. Patients with an extent of fibrosis ≥20% as per an HRCT of the chest performed within 12 months prior to Visit 1 or during the screening period (if not available) and confirmed by central review.
7. Patients with a Forced vital capacity (FVC) ≥45% predicted at Visit 1. Predicted normal values will be calculated according to Global Lung Initiative (GLI).
8. Patients with haemoglobin-corrected diffusing capacity of the lungs for carbon monoxide (DLCO) ≥20% predicted at Visit 1.

Further inclusion criteria apply.

Exclusion criteria:

1. Acute exacerbation of IPF within at least 12 weeks prior to Visit 1 and/or during the screening period (investigator-determined).
2. Relevant airways obstruction (pre-bronchodilator forced expiratory volume in 1 second (FEV1)/FVC <0.7) at Visit 1.
3. Lower respiratory tract infection requiring treatment within 4 weeks prior to Visit 1 and/or during the screening period.
4. Significant PH defined by any of the following:

   * Previous clinical or echocardiographic evidence of significant right heart failure according to investigator's judgement
   * History of right heart catheterisation showing a cardiac index ≤2 L/min/m^²
   * PH requiring parenteral therapy with prostanoids
5. On nintedanib or pirfenidone treatment for less than 12 weeks prior Visit 1, planning to start nintedanib or pirfenidone within the first 12 weeks of investigational medicinal product (IMP) treatment or on combined nintedanib plus pirfenidone treatment. Newly diagnosed patients considered in need of SoC treatment by the treating physician, who would be withheld SoC treatment only for the sake of participation in the trial, should also be excluded.
6. Cardiovascular comorbidities including

   * Severe hypertension (uncontrolled under treatment≥160/100 mmHg at multiple occasions) within 3 months of Visit 1
   * Myocardial infarction, stroke, or transient ischemic attack within 6 months of Visit 1
   * Unstable cardiac angina within 6 months of Visit 1
7. Life expectancy for any concomitant disease other than IPF <2.5 years (investigator assessment).

Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in FVC (mL) at 12 weeks | Baseline, 12 weeks

SECONDARY OUTCOMES:
Absolute change from baseline in log 10- transformed SP-D plasma concentration at 12 weeks | Baseline, 12 weeks
  SP-D=Surfactant protein D
Absolute change from baseline in distance walked (m) during 6MWT at 12 weeks | Baseline, 12 weeks
  6MWT=6-minute walk test
Absolute change from baseline in FVC % predicted at 12 weeks | Baseline, 12 weeks
Absolute change from baseline in DLCO % predicted at 12 weeks | Baseline, 12 weeks
  DLCO=Diffusing Capacity of the Lungs for Carbon Monoxide
Absolute change from baseline in SpO2 on room air at rest at 12 weeks | Baseline, 12 weeks
  SPO2=Oxygen saturation

CONTACTS AND LOCATIONS:
Locations (49):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner - University Medical Center Tucson, Tucson, Arizona
  - University of Florida, Gainesville, Florida
  - Renstar Medical Research, Ocala, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - University of Missouri Health System, Columbia, Missouri
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Clinical Trials Center of Middle Tennessee, LLC, Franklin, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia
- Australia (3):
  - The Prince Charles Hospital, Chermside, Queensland
  - Monash Health, Clayton, Victoria
  - Institute for Respiratory Health, Nedlands, Western Australia
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Canada (4):
  - Synergy Respiratory Care, Sherwood Park, Alberta
  - Kelowna Respirology & Allergy Research, Kelowna, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- Germany (2):
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Medizinische Hochschule Hannover, Hanover
- Italy (5):
  - ASST Papa Giovanni XXIII, Bergamo
  - A. O. Universitaria Careggi, Florence
  - A.O. dei Colli, Napoli
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Azienda Ospedaliera Universitaria Citta Della Salute E Della Scienza Di Torino, Torino
- Japan (6):
  - Tosei General Hospital, Aichi, Seto
  - University of Fukui Hospital, Fukui, Yoshida-gun
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
- South Korea (4):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Inje University Haeundae Paik Hospital, Busan
  - Soonchunhyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Vall Hebron, Barcelona
  - Hospital Universitari de Bellvitge, L Hospitalet Del Llobregat
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Virgen del Rocío, Seville
- Cantonal Hospital of Aarau, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor'spublication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com